CLINICAL TRIAL: NCT01254656
Title: A Long Term Open-Label Extension Study Of Lersivirine For The Treatment Of HIV-1 Infection
Brief Title: A Long Term Safety Study Of Lersivirine For The Treatment Of HIV-1 Infection In Subjects Who Have Completed Treatment With Lersivirine In Studies A5271015 And A5271022
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5271037
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-01

CONDITIONS: HIV-1
MeSH Terms: interventions — UK 453,061; efavirenz; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- LRV 500mg (Experimental)
  Interventions: Drug: lersivirine
- LRV 750mg +TVD (Experimental)
  Interventions: Drug: lersivirine
- EFV (Active Comparator)
  Interventions: Drug: efavirenz
- LRV 750mg+ DRV/r + OBT (Experimental)
  Interventions: Drug: lersivirine
- LRV 1000mg +DRV/r + OBT (Experimental)
  Interventions: Drug: lersivirine
- ETR (Active Comparator)
  Interventions: Drug: etravirine

INTERVENTIONS:
Drug: lersivirine — Lersivirine 500 mg tablets PO taken once daily + tenofovir DF 300 mg/emtricitabine 200 mg tablets PO once daily
  Arms: LRV 500mg
Drug: lersivirine — Lersivirine 750 mg tablets PO taken once daily + tenofovir DF 300 mg/emtricitabine 200 mg tablets PO once daily
  Arms: LRV 750mg +TVD
Drug: efavirenz — Efavirenz 600 mg tablets PO taken once daily + tenofovir DF 300 mg/emtricitabine 200 mg tablets PO once daily
  Arms: EFV
Drug: lersivirine — Lersivirine 750 mg tablets PO taken once daily + darunavir 600 mg tablets/ritonavir 100 mg tablets or capsules PO taken twice daily + 1 optimized NRTI
  Arms: LRV 750mg+ DRV/r + OBT
Drug: lersivirine — Lersivirine 1000 mg PO tablets + darunavir 600 mg tablets/ritonavir 100 mg tablets or capsules PO taken twice daily + 1 optimized NRTI
  Arms: LRV 1000mg +DRV/r + OBT
Drug: etravirine — Etravirine 200 mg PO tablets + darunavir 600 mg tablets/ritonavir 100 mg tablets or capsules taken twice daily + 1 optimized NRTI
  Arms: ETR

SUMMARY:
This is a study to assess long-term safety and efficacy of lersivirine in patients who have completed 96 weeks of treatment with lersivirine in studies A5271015 and A5271022.

DETAILED DESCRIPTION:
The trial was terminated prematurely on January 29, 2013, due to the decision of the sponsor to discontinue development of lersivirine. The decision to terminate the trial was not based on any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Patients must complete of 96 weeks of treatment with lersivirine (or comparator where required by local regulation) in one of the parent protocols (A5271015 or A5271022).
* Patients must have had a viral load less than 50 copies/mL at Week 84 of the parent protocol.
* For women who can have children, a negative urine pregnancy test at the Day 1 visit.

Exclusion Criteria:

* Patients with any Grade 4 Division of AIDS toxicity (except for lipids and asymptomatic glucose elevations will not be included in this trial.
* Patients being treated with another investigational product or in another clinical trial, except the lersivirine parent protocols will not be included in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Australia (2):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Melbourne, Victoria
- Pfizer Investigational Site, Nova Iguaçu, Rio de Janeiro, Brazil
- Canada (2):
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Italy (2):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Torino
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico
- Poland (2):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Warsaw
- South Africa (6):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Soweto, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Cape Town, Western Cape
  - Pfizer Investigational Site, Pretoria
- Switzerland (3):
  - Pfizer Investigational Site, Lugano
  - Pfizer Investigational Site, Sankt Gallen
  - Pfizer Investigational Site, Zurich
- United Kingdom (2):
  - Pfizer Investigational Site, Brighton, East Sussex
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271037&StudyName=A%20Long%20Term%20Safety%20Study%20Of%20Lersivirine%20For%20The%20Treatment%20Of%20HIV-1%20Infection%20In%20Subjects%20Who%20Have%20Completed%20Treatment%20With%20Lersivirine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had completed 96 weeks of treatment with lersivirine in the A5271015 parent study were enrolled in this extension study. One participant from a second parent study (A5271022) was initially enrolled in Study A5271037, but later discontinued from A5271037.
Pre-assignment Details: Participants were required to have plasma HIV-1 ribonucleic acid (RNA) <50 copies/mL at Week 84 of the parent protocol. Of 108 participants screened in the parent protocol A5271015, 47, 43, and 18 participants from the lersivirine 500 mg, lersivirine 750 mg, and efavirenz 600 mg groups, respectively, were enrolled in Study A5271037.
Groups:
- Lersivirine (LRV) 500 mg: Participants received LRV 500 mg orally once daily (QD). In addition participants received treatment with tenofovir disoproxil fumarate (TDF) 300 mg/emtricitabine (FTC) 200 mg orally QD
- LRV 750 mg: Participants received LRV 750 mg orally QD. In addition participants received treatment with tenofovir disoproxil fumarate (TDF) 300 mg/emtricitabine (FTC) 200 mg orally QD
- Efavirenz (EFV) 600 mg: Participants received EFV 600 mg orally QD. In addition participants received treatment with tenofovir disoproxil fumarate (TDF) 300 mg/emtricitabine (FTC) 200 mg orally QD
Period: Overall Study
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Started | 47 | 43 | 18
Treated | 47 | 43 | 18
Completed | 0 | 0 | 0
Not Completed | 47 | 43 | 18
Not completed — Discontinued due to termination of study | 40 | 39 | 13
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg | Total
Number analyzed (Participants) | 47 | 43 | 18 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (8.4) | 35.8 (8.7) | 38.5 (7.8) | 36.6 (8.4)
Age, Customized [Number; unit: Participants]
  < 18 Years | 0 | 0 | 0 | 0
  18 - 44 Years | 41 | 37 | 14 | 92
  45 - 64 Years | 6 | 6 | 4 | 16
  >= 65 Years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 8 | 29
  Male | 37 | 32 | 10 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma Human Immunodeficiency Virus - 1 (HIV-1) Ribonucleic Acid (RNA) Level <50 Copies/mL at 144 Weeks From Day 1 of the Parent Protocol
Description: Number of participants with HIV-1 RNA level <50 copies/mL plasma was summarized at 48 weeks i.e. 144 weeks from Day 1 of the parent protocol. Roche Amplicor HIV-1 Monitor assay was used to measure the HIV-1 RNA level.
Time Frame: 144 Weeks from Day 1 of the parent protocol
Population: All participants enrolled in this protocol constituted the analysis population associated with each of the parent protocols and all available data were used for efficacy analyses.
Measure: Number; unit: Participants
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Number analyzed (Participants) | 47 | 43 | 18
Participants | 40 | 40 | 16

2. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA Level <50 Copies/mL up to Week 208
Description: Number of participants with HIV-1 RNA level <50 copies/mL plasma was summarized at last visit. Abbott RealTime HIV-1 assay was used to measure the HIV-1 RNA level.
Time Frame: Up to Week 208
Population: Analyses included all enrolled participants. Last visit used the last available visit of each participant. Discontinued from study, lost to follow-up, or missing HIV-1 RNA level data at last visit were considered to have HIV-1 RNA levels >=50 copies/mL. Participants discontinued due to program termination were not considered as discontinuations.
Measure: Number; unit: Participants
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Number analyzed (Participants) | 47 | 43 | 18
Participants | 39 | 38 | 13

3. Secondary Outcome: Change From Baseline in CD4+ Lymphocyte Counts (Absolute) at 144 Weeks From Day 1 of the Parent Protocol
Description: Participant's immunological status assessed by CD4+ lymphocyte count (absolute and percentage) at 48 weeks (ie, 144 weeks from Day 1 of the parent protocol)
Time Frame: 144 Weeks from Day 1 of the parent protocol
Population: All participants enrolled in this protocol constituted the analysis population associated with each of the parent protocols and all available data were used for efficacy analyses. Last observation carried forward (LOCF) was used to impute missing values.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Number analyzed (Participants) | 47 | 43 | 18
cells/uL | 293 (206) | 302 (163) | 303 (163)

4. Secondary Outcome: Change From Baseline in CD4+ Lymphocyte Counts (Percentage) at 144 Weeks From Day 1 of the Parent Protocol
Description: as for outcome 3
Time Frame: 144 Weeks from Day 1 of the parent protocol
Population: All participants enrolled in this protocol constituted the analysis population associated with each of the parent protocols and all available data were used for efficacy analyses. LOCF was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Number analyzed (Participants) | 47 | 43 | 18
Percentage | 13 (6) | 13 (5) | 13 (6)

5. Secondary Outcome: Change From Baseline in CD4+ Lymphocyte Counts (Absolute) at 192 Weeks From Day 1 of the Parent Protocol
Description: Participant's immunological status assessed by CD4+ lymphocyte count (absolute and percentage) at 192 weeks from Day 1 of the parent protocol.
Time Frame: 192 Weeks from Day 1 of the parent protocol
Population: Analyses included all enrolled participants. Week 192 data are presented, as Week 208 had few participants. For participants who discontinued prematurely, LOCF was used to impute values for post discontinuation visits. Participants who discontinued due to termination of the program were not included in the analysis for the post termination visits.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Number analyzed (Participants) | 38 | 34 | 18
cells/uL | 308 (191) | 304 (159) | 300 (220)

6. Secondary Outcome: Change From Baseline in CD4+ Lymphocyte Counts (Percentage) at 192 Weeks From Day 1 of the Parent Protocol
Description: as for outcome 5
Time Frame: 192 Weeks from Day 1 of the parent protocol
Population: Analyses included all enrolled participants. Week 192 data are presented as Week 208 had few participants. For participants who discontinued prematurely, LOCF was used to impute values for post discontinuation visits. Participants who discontinued due to termination of the program were not included in the analysis for the post termination visits.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Number analyzed (Participants) | 38 | 34 | 18
Percentage | 13 (6) | 15 (6) | 12 (6)

7. Secondary Outcome: Virology Analysis Participant Accountability From Week 96 Through Study Termination
Description: Virology analysis included virus susceptibility (phenotype and genotype)to a standard panel of approved antiretrovirals as determined by the Monogram Biosciences PhenoSense GT assay. Below analysis table included the following parameters: 1. "protocol-defined treatment failure" was defined as an increase in HIV-1 RNA to detectable levels (≥50 copies/mL) on 2 consecutive measurements, the second measurement taken no more than 14 days after the first measurement); 2. "Treatment failure": treatment failure (both virologic and non-virologic) was defined as a subject who met the protocol-defined treatment failure criterion or discontinued from the study; 3. "NRTI or NNRTI resistance mutations": nucleoside reverse transcriptase inhibitor or lersivirine-associated resistance-associated mutations (RAM) based on the International AIDS Society-USA (IAS-USA) RAM guidelines; 4. 'with result' meant an analyzed sample returned genotypic result or phenotypic result or both.
Time Frame: Week 96 through study termination
Population: The virology analysis set included only evaluable participants i.e. those having samples with valid genotypic or phenotypic susceptibility testing results and HIV-1 RNA >500 copies/mL. However, samples with observed emergence of resistance-associated mutations and HIV-1 RNA level ≤500 copies/mL or missing HIV-1 RNA level, were also noted.
Measure: Number; unit: Participants
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Number analyzed (Participants) | 47 | 43 | 18
Participants
  Treatment failure (TF) | 8 | 5 | 5
  Protocol defined treatment failure | 4 | 3 | 0
  TF analysed - HIV-1 RNA >500 c/mL | 1 | 0 | 0
  TF analysed - HIV-1 RNA >500 c/mL with result | 1 | 0 | 0
  TF analysed - HIV-1 RNA <= 500 c/mL | 5 | 2 | 2
  TF analysed - HIV-1 RNA <= 500 c/mL with result | 2 | 1 | 0
  NRTI or NNRTI resistance mutations | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 208
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. Treatment emergent AEs included new treatment emergent AEs in A5271037 as well as AEs that were ongoing at the time of enrolment in A5271037 and had a worsened severity grading from that reported in A5271015. All causality events were reported.
Arm/Group | Lersivirine (LRV) 500 mg | LRV 750 mg | Efavirenz (EFV) 600 mg
Serious Adverse Events (participants affected / at risk) | 6/47 | 5/43 | 0/18
Other Adverse Events (participants affected / at risk) | 30/47 | 35/43 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lersivirine (LRV) 500 mg (N=47) | LRV 750 mg (N=43) | Efavirenz (EFV) 600 mg (N=18)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Syphilis (Infections and infestations) | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lersivirine (LRV) 500 mg (N=47) | LRV 750 mg (N=43) | Efavirenz (EFV) 600 mg (N=18)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Ocular toxicity (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 3 | 0
Discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Nodule (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Anal chlamydia infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Chlamydial infection (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Gonorrhoea (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 1
Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 1 | 1
Oropharyngeal gonococcal infection (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 4 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0
Proctitis gonococcal (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Syphilis (Infections and infestations) | 1 | 0 | 1
Tinea barbae (Infections and infestations) | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3
Urethritis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Blood cholesterol increased (Investigations) | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase abnormal (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Lipids increased (Investigations) | 1 | 0 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0
Parasitic test positive (Investigations) | 0 | 1 | 0
Simplex virus test positive (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Areflexia (Nervous system disorders) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Genital lesion (Reproductive system and breast disorders) | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Perineal erythema (Reproductive system and breast disorders) | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular microlithiasis (Reproductive system and breast disorders) | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Spider vein (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated on 29 Jan 13 due to termination of lersivirine development program. All participants were enrolled from study A5271015 except one from A5271022. Above summarized outcome measures included participants enrolled from A5271015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.